CLINICAL TRIAL: NCT06653673
Title: ChatGPT-Supported Online Group-Guided Self-Help Program
Brief Title: The Effect of a ChatGPT-Supported Online Group-Guided Self-Help Program on Uncontrolled and Emotional Eating Behaviors and Body Image in Overweight and Obese Woman Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülsüm Zekiye Tuncer, Assistant Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9128-GOA
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Overweight (BMI > 25); Obesity and Overweight; Emotional Eating; Binge Eating
Keywords: ChatGPT; Self Help; group; online
MeSH Terms: conditions — Overweight; Obesity; Emotional Eating; Bulimia

STUDY DESIGN:
Intervention Model Description: This study is planned to be conducted as a Randomized Controlled Trial (RCT).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChatGPT supported Online Guided Self-Help Program (GSHP) (Experimental): The experimental group will participate in the ChatGPT-supported Online Group Guided Self-Help Program.
  Interventions: Behavioral: ChatGPT supported Online Guided Self-Help Program (GSHP)
- Control group (No Intervention): The control group will consist of participants placed on a waitlist.

INTERVENTIONS:
Behavioral: ChatGPT supported Online Guided Self-Help Program (GSHP) — Guided Self-Help Program (GSHP)
  The Guided Self-Help Program (GSHP) was developed by Fairburn and Carter for patients with binge eating disorder and later adapted to address various eating behaviors, forming an intervention protocol. GSHP modules consist of:
  Starting self-monitoring, Establishing regular eating patterns, Applying the "mindful eating" rule and developing alternatives to emotional eating, Practicing problem-solving exercises, Addressing diet-related issues and body image, and Termination modules.
  Session Structure:
  Session 1 focuses on tracking eating patterns and raising self-awareness about eating habits. Individuals are asked to maintain a daily record via a shared Google Forms link. This food diary is later processed through ChatGPT, and personalized feedback is provided.
  Session 2 provides psychoeducation on developing regular eating patterns. It emphasizes recognizing hunger and satiety cycles and reducing triggers. Participants are asked to log their meals daily
  Arms: ChatGPT supported Online Guided Self-Help Program (GSHP)

SUMMARY:
Nurses with overweight and female gender characteristics often experience disruptions in their eating behaviors due to stressful working conditions. These disruptions can lead to physical and psychosocial problems (Nicholls et al., 2017). Studies have shown that guided self-help programs, based on cognitive behavioral therapy interventions, are effective in addressing uncontrolled and emotional eating behaviors (Carrard et al., 2011; Cachelin et al., 2015). However, the use of supportive tools to assist the facilitator in group-based interventions of these evidence-based self-help programs and their impact on individual recovery processes remain unexplored. Additionally, no studies have been found investigating the application of these AI-supported guided self-help programs among female nurses, who are frequently exposed to stress and at high risk of obesity.

Given the demanding workloads of nurses, cost-effective and easily accessible online programs have been found to promote recovery (Jenkins et al., 2021). Therefore, it is essential to test this AI-supported program in an online group format with overweight and obese woman nurses.

The aim of this study is to evaluate the effect of a ChatGPT-supported online group-guided self-help program on uncontrolled and emotional eating behaviors and body image in overweight and obese woman nurses through a randomized controlled trial. Participants will be recruited via an announcement shared on social media platforms (Instagram). Nurses who respond to the announcement will be asked to complete a survey through Google Forms. Those randomly assigned to the intervention group will participate in online group sessions conducted via Google Meets. Pre- and post-test data will be collected using Google Forms.

ELIGIBILITY:
Inclusion Criteria:

* Hold at least a bachelor's degree in nursing from a nursing school.
* Work as a nurse in an institution.
* Be a woman.
* Have a BMI (Body Mass Index) greater than 24.99.
* Not have a hearing impairment that would prevent them from understanding and completing verbal instructions.
* Have access to a smartphone or computer with a camera.
* Agree to participate in the study.
* Score 50 or higher on the emotional eating and external eating subscales of the Dutch Eating Behavior Questionnaire (DEBQ).

Exclusion Criteria:

* Refusal to participate in the study.
* Diagnosis of chronic diseases such as diabetes, hyperlipidemia, hypertension, or hyperthyroidism.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — woman participant
Enrollment: 44 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Dutch Eating Behavior Questionnaire (DEBQ) | 8 weeks
  The Dutch Eating Behavior Questionnaire (DEBQ) was developed by Van Strien, Frijters, Jan, Bergers, and Defares (1986) to measure emotional, external, and restrained eating behaviors. The questionnaire consists of 33 items divided into three subscales:
  Restrained Eating (10 items) - Example: "Do you deliberately eat foods that are slimming?" Emotional Eating (13 items) - Example: "Do you have a desire to eat when someone upsets you?" External Eating (10 items) - Example: "Do you feel like eating when you pass by a café or snack bar?" Each item is rated on a 5-point Likert scale (1 = Never, 5 = Very often). The 31st item is reverse-scored.
  The psychometric properties of the DEBQ were validated in Turkish by Bozan, Baş, and Aşçı (2011), confirming the original three-factor structure. In their study, the Cronbach's alpha coefficients for the subscales were found to be:
  Emotional Eating: .90 Restrained Eating: .94 External Eating: .96 These reliability values indicate high internal con

CONTACTS AND LOCATIONS:
Overall Officials: Gülsüm Zekiye TUNCER, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University Faculty of Nursing, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In our ethics approval, it is stated that participant data confidentiality will be ensured. The ethical approval has been obtained in this manner.